CLINICAL TRIAL: NCT04217473
Title: A Phase 1, Open-Label, Dose-Escalation Clinical Trial of Tumor Necrosis Factor Alpha and Interleukin 2 Coding Oncolytic Adenovirus TILT-123 in Melanoma Patients Receiving Adoptive Cell Therapy With Tumor Infiltrating Lymphocytes
Brief Title: TNFalpha and Interleukin 2 Coding Oncolytic Adenovirus TILT-123 During TIL Treatment of Advanced Melanoma
Acronym: TUNINTIL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TILT Biotherapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILT-T215
Record Dates: First submitted 2019-12-19; First posted 2020-01-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Melanoma
Keywords: oncolytic virus; T-cell therapy; immunotherapy; TILT
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: open-label, single arm, dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TILT-123 (Experimental): Patients will receive administrations of TILT-123. Patients will also receive Tumor Infiltrating Lymphocytes (TILs) during the treatment phase.
  Escalation to the next dose of TILT-123 level will occur when the safety data has been evaluated for all patients in the preceding dose level.
  Interventions: Biological: TILT-123

INTERVENTIONS:
Biological: TILT-123 — TNFalpha and IL-2 coding oncolytic adenovirus TILT-123

SUMMARY:
This is an open-label, phase 1, first-in-human (FIH), dose-escalation, multicenter, multinational trial evaluating the safety of oncolytic adenovirus TILT-123 as monotherapy and in association with T-cell therapy with TILs in metastatic melanoma patients.

DETAILED DESCRIPTION:
The primary objective of the trial is to evaluate the safety of TILT-123. The approach has the potential to a) increase the efficacy of adoptive T-cell therapy, b) remove the need for toxic pre- and post-conditioning regimens, c) yield the combined anti-tumor benefits of armed oncolytic viruses and T-cell therapy.

Dose escalation of TILT-123 injection will take place between cohorts not intra-patient and will be determined based on Dose Limiting Toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent before any trial-related activities.
* Male or female, between 18-75 years of age (both included).
* Pathologically confirmed previously treated refractory or recurrent stage 3-4 melanoma, which cannot be treated with curative intent with available therapies.
* At least one prior line of medical treatment is required (for example checkpoint inhibitors, kinase inhibitors, interleukin-2). Multiple prior therapies (e.g. surgery, checkpoint inhibitors, kinase inhibitors, interleukin-2, interferon, chemotherapy, radiation) are allowed.
* A > 9 mm tumor (in diameter, typically a minimum of 1 cm3 in volume) without signs of necrosis must be available for biopsy/operation to enable growing of TILs.
* At least one additional tumor (>14 mm in diameter) must be available for injections and biopsies for correlative analyses. The disease burden must be measurable, but does not need to fulfil RECIST 1.1.
* Eligible for adoptive T-cell therapy with tumor infiltrating lymphocytes

Adequate hepatic, cardiac and renal functions as following:

1. Platelets > 75 000/mm3
2. Haemoglobin ≥ 100 g/L.
3. AST and ALT < 3 x ULN.
4. GFR >60 ml/min (Cockcroft-Gault formula).
5. Leukocytes (WBC) > 3,0
6. Bilirubin <1.5 x ULN

   * Men and women must be willing to use adequate forms of contraception from screening, during the trial, and for a minimum of 90 days after end of treatment, in accordance with the following:
   * Women of childbearing potential: Barrier contraceptive method (i.e. condom) must be used in addition to one of the following methods: Intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections).
   * Women not of childbearing potential: Barrier contraceptive method (i.e. condom) must be used.
   * Men: Barrier contraceptive method (i.e. condom) must be used.
   * Demonstrated WHO performance score of 0-1 at screening.
   * Life expectancy time longer than 3 months.
   * Capable of understanding and complying with parameters as outlined in the protocol.
   * BRAF negative or positive.

Exclusion Criteria:

* Use of immunosuppressive medications (corticosteroids or drugs used in treatment of autoimmune disease). Exempted are the following which can be allowed at screening and during the trial: replacement corticosteroids if e.g. the patient has adrenal insufficiency after prior immunotherapy; pulmonal and topical treatments; up to 20 mg of prednisone/prednisolone.
* History of another active invasive cancer as judged by the investigator within the past 3 years except basalioma.
* Treated with any anti-cancer therapy for melanoma 30 days prior to enrolment. Anti-cancer therapy for melanoma is defined as anti-cancer agents (immunotherapy, signal-transduction inhibitors [e.g. BRAF and MEK inhibitors], cytotoxic chemotherapy), radiotherapy and investigational agents. An investigational agent is any drug or therapy that is currently not approved for use in humans.
* Uncontrolled cardiac or vascular diseases.
* History of heart attack or cerebral stroke within the previous 12 months before screening or is not recovered from an older heart attack or cerebral stroke.
* LDH value > 3 x ULN.
* History of hepatic dysfunction, hepatitis or HIV.
* History of coagulation disorder.
* Any other disease which prevent participation in the opinion of the investigator.
* Female patients who are pregnant, breastfeeding or intends to become pregnant.
* Untreated brain metastases. Treated brain metastases which have not progressed in 3 months prior to screening are allowed.
* Previously treated with any oncolytic adenovirus that was administered intratumorally.
* Previously treated with adoptive cell therapy.
* Allergy to TILT-123, TIL, or ingredients present in the investigational medicinal products.
* Administered an investigational medicinal product or device in another clinical trial within 30 days prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with any (serious and non-serious) Adverse Events prior to TIL administration. | 36 days
Number of Participants with abnormal laboratory values prior to TIL administration. | 36 days
Number of Participants with vital sign abnormalities prior to TIL administration. | 36 days
Safety assessed by 12- lead electrocardiograms (ECGs) Adverse Events prior to TIL administration. | 36 days
  Any clinically significant adverse changes on the ECG will be reported as Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Principal Investigator — CCIT, Herlev Hospital, Copenhagen University; Brigitte Dréno, Principal Investigator — CHU Nantes, Nantes University Hospital
Locations (2):
- National Center for Cancer Immune Therapy Herlev Hospital, Copenhagen University, Copenhagen, Denmark
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clubb JHA, Pakola SA, Joenvaara S, Kudling TV, Tohmola T, Arias V, Jirovec E, van der Heijden M, Quixabeira DCA, Pasanen A, Haybout L, Ojala N, Basnet S, Eleuteri A, Ferrero JD, Hirvenoja S, Svane IM, Maenpaa J, Jalkanen K, Block MS, Alanko T, Monberg T, Zahraoui S, Gronberg-Vaha-Koskela S, Salmelin N, Kistler C, Havunen R, Sorsa S, Manuel Dos Santos J, Cervera-Carrascon V, Kanerva A, Hemminki O, Renkonen R, Hemminki A. Dyslipidemia-associated natural IgM improves oncolytic virus TILT-123 efficacy through antibody-dependent enhancement in solid tumors. Mol Ther. 2026 Jan 20:S1525-0016(26)00020-1. doi: 10.1016/j.ymthe.2026.01.019. Online ahead of print. PMID 41566775
- [Derived] Jirovec E, Quixabeira DCA, Clubb JHA, Pakola SA, Kudling T, Arias V, Haybout L, Jalkanen K, Alanko T, Monberg T, Khammari A, Dreno B, Svane IM, Block MS, Adamo DA, Maenpaa J, Kistler C, Sorsa S, Hemminki O, Kanerva A, Santos JM, Cervera-Carrascon V, Hemminki A. Single intravenous administration of oncolytic adenovirus TILT-123 results in systemic tumor transduction and immune response in patients with advanced solid tumors. J Exp Clin Cancer Res. 2024 Nov 6;43(1):297. doi: 10.1186/s13046-024-03219-0. PMID 39506856
- [Derived] Havunen R, Kalliokoski R, Siurala M, Sorsa S, Santos JM, Cervera-Carrascon V, Anttila M, Hemminki A. Cytokine-Coding Oncolytic Adenovirus TILT-123 Is Safe, Selective, and Effective as a Single Agent and in Combination with Immune Checkpoint Inhibitor Anti-PD-1. Cells. 2021 Jan 27;10(2):246. doi: 10.3390/cells10020246. PMID 33513935
- [Derived] Cervera-Carrascon V, Quixabeira DCA, Havunen R, Santos JM, Kutvonen E, Clubb JHA, Siurala M, Heinio C, Zafar S, Koivula T, Lumen D, Vaha M, Garcia-Horsman A, Airaksinen AJ, Sorsa S, Anttila M, Hukkanen V, Kanerva A, Hemminki A. Comparison of Clinically Relevant Oncolytic Virus Platforms for Enhancing T Cell Therapy of Solid Tumors. Mol Ther Oncolytics. 2020 Mar 19;17:47-60. doi: 10.1016/j.omto.2020.03.003. eCollection 2020 Jun 26. PMID 32322662